CLINICAL TRIAL: NCT01756872
Title: Determining the Accuracy of Clinical Measures of Ovarian Reserve in Predicting Successful In Vitro Fertilisation (IVF)Treatment.
Brief Title: Clinical Measures of Ovarian Reserve in Predicting IVF Success
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Oxford Fertility Unit (Other)
Responsible Party: Sponsor
Other Study IDs: NDOG-12/SC/0277
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Infertility, Female
Keywords: infertility; Assisted reproductive technology; ovarian reserve
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ovarian reserve study participants: Measurements of ovarian reserve for women attending the Oxford Fertility Unit having their first IVF/IVF-ICSI cycle.
  Interventions: Procedure: Measurements of ovarian reserve

INTERVENTIONS:
Procedure: Measurements of ovarian reserve — Blood test (AMH, E2, FSH) Ultrasound measurement of antral follicle count and ovarian volume

SUMMARY:
The purpose of this study is to find out more about tests used to estimate the number of eggs a woman has remaining in her ovaries (her 'ovarian reserve'). It is thought that women who have a greater number of eggs or ovarian reserve may have a better chance of successful in vitro Fertilisation (IVF) treatment than those who have a smaller number of eggs. Accurately predicting the likely outcomes of IVF would be of great benefit for counselling patients before they go through expensive and demanding treatments such as IVF and IVF with Intracytoplasmic sperm injection (IVFICSI).

Over the past two decades, many endocrine and ultrasound markers have been designed and are now used as indicators of ovarian reserve. A number of screening tests are utilized to measure these markers, either by ultrasound scanning techniques or taking blood samples. However it is not yet known which, if any, best predict the outcome of IVF treatment. We would like to investigate these various measures of ovarian reserve to determine which are most accurate, particularly for predicting live birth rates, as up to now only poor to moderate quality evidence has been available for this outcome.

This will be a prospective cohort study of 300 women who already intend to undergo IVF/IVF-ICSI treatment. Study participants will have one extra blood sample and ultrasound examination, for the purposes of measuring markers of their ovarian reserve, at the start of their IVF/IVFICSI treatment cycle. No other interventions will be required and their treatment cycle will not be affected by their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Female, aged 18 years or above.
* First cycle of ovarian stimulation.
* Suitable for standard 'long protocol' IVF/IVF-ICSI cycle.

Exclusion Criteria:

* The participant does not understand the English language, or has special communication needs. This is because it is impractical to provide, for this small scale study, information sheets and consent forms in other languages except English.
* Patients unsuitable for standard 'long protocol' IVF/IVFICSI cycle

  * Presence of endometrioma or any other kind of ovarian cyst > 20mm diameter.
  * Presence of Polycystic Ovarian Syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women attending the Oxford Fertility Unit planning an IVF/IVF-ICSI treatment cycle
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Live birth rate per cycle | up to one year after last appointment of final participant

CONTACTS AND LOCATIONS:
Overall Officials: Tim Child, Principal Investigator — University of Oxford
Locations (1):
- Oxford Fertility Unit, Oxford, United Kingdom